CLINICAL TRIAL: NCT00321126
Title: Effect of Zinc Supplementation on the Immune and Inflammatory Responses of Children to Shigella Flexneri Infection, and Correlation With Clinical Severity of Illness and Growth Following recoveryEffect of Zinc Supplementation on the Immune and Inflammatory Responses of Children to Shigella Flexneri Infection, and Correlation With Clinical Severity of Illness and Growth Following Recovery
Brief Title: Zinc Supplementation in Shigella Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Karolinska Institutet (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 97-020
Record Dates: First submitted 2006-05-02; First posted 2006-05-03 (Estimated); Last update posted 2006-05-03 (Estimated); Status verified 2006-05

CONDITIONS: Testing Effect of Intervention
Keywords: Zinc; Shigella; Children; Bangladesh
MeSH Terms: conditions — Dysentery, Bacillary

INTERVENTIONS:
Drug: Children in the zinc group received 20 mg of elemental zinc as acetate per day in a twice-daily dose for two weeks.

SUMMARY:
Shigellosis is a major cause of morbidity and mortality in young children in Bangladesh and other developing countries. Further, the increasing emergence of resistance to a wide range of antibiotics is of great concern. Another major public health problem in Bangladesh is malnutrition, which is closely linked with shigellosis and with a high mortality. In Shigellosis, a heavy nutritional burden is placed on children and vital micronutrients such as vitamin A is lost in the urine. We recently found that the immune response in S. Flexneri infection was lower in children who were severely malnourished (weight-for-age≤65% as a percentage of the National Centre for Health Statistics median) when compared to children with weight-for-age from >65-75%. T cell responses were primarily affected with lowered CD4/CD8 ratios, lowered proliferative responses to T cell mitogens, Conconavalin A (ConA) and phytohaemagglutinin (PHA). However, proliferation of pheripheral blood mononuclear cells (PBMs) was lowered only in the presence of autologous plasma suggesting that a factor(s) in plasma, probably nutritional, rather than a defect in cells themselves was responsible. In children with S. dysenteriae 1 infection, proliferative responses to PHA were similarly lowered in the presence of autologous plasma but inhibition correlated to lowered transferring levels in plasma and not to the weight-for-age of the children. Also severely malnourished children with either S. flexneri or S. dysenteriae 1 infection were more severely ill. These findingings show that immunity in malnourishrd children with shigella infection is impaired which may lead to more severe illness. As zinc has profound effects on immunity as well as clinical outcome in diarrhoeal diseases, it is possible that zinc deficiency may be a factor in reducing immunity and increasing severity of acute illness in malnourished children with shigellosis. In this study, we will investigate the effect of zinc supplementation, in a double blind placebo controlled trial, on inflammatory responses, outcome of acute illness and growth following recovery from acute illness with S. flexneri infection.

DETAILED DESCRIPTION:
Study design: The study was a double blind randomised clinical trial using zinc and placebo using multivitamin base.Study subjects: Fifty six children of both sex aged between 12-59 months were studied in the study ward who attended the Dhaka Hospital of International Centre for Diarrhoeal Disease Research, Bangladesh with shigellosis. The patients were initially screened for the study. Stool samples were examined microscopically and stool was cultured for enteric bacterial pathogens. Children whose stool cultures were positive for shigella species were included in the study. Selection of the patients were based on the following criteria: age between 12-59 months, moderate malnutrition (61-75% Weight / Age - NCHS Median), duration of diarrhoea of 5 days, and culture confirmed shigella spp in stool on enrolment. Measurements of weight and length (height) were performed by using the WHO Manual28. The exclusion criteria were as follows: measles infection in the past six months; presence of obvious systemic illnesses, such as pneumonia, meningitis, septicaemia, leukemoid reaction, haemolytic uremic syndrome etc; zinc supplementation; severe malnutrition; residence in a location requiring a journey of > 2 hour from the Dhaka Hospital of the ICDDR,B ; and refusal to give consent. Signed informed consent was obtained from the guardian of each paediatric patients before enrolment according to the guidelines of the ethical review committee of the ICDDR,B. The study was conducted between January 1999 -December 2002.Study Groups: There were two study groups, one received zinc acetate with multivitamin syrup and antibiotic i.e. pivmecillinum and the other with placebo and pivmecillinum . Composition of syrup: For both groups, the base syrup or multivitamin syrup was of the same composition. In addition to this, zinc acetate (20 mg elemental Zn/ 5 ml) was mixed in the multivitamin syrup for the zinc supplemented group to receive 20 mg elemental zinc per day.Composition of base/ multivitamin syrup: Every 5 ml of the multivitamin syrup contained the following: vitamin A (3000IU), vitamin D (600 IU), thiamin (1.2 mg), riboflavin (2.0 mg), nicotinamide (6.0 mg) and calcium pantothanate (6 mg).Dose of zinc: Subjects of zinc group received 20 mg elemental zinc as acetate per day in a twice-daily dose for a period of 2 weeks. Methods: A block randomization procedure was performed by using a random table to assign a equal number of patients to the zinc supplemented and placebo group. Twenty eight in each group were allocated to zinc or placebo using block randomization. Double blinding was done by having identical coloured bottles of syrup labeled with serial numbers, which were allocated to the children of the 2 groups chronologically. The zinc syrup containing zinc and the multivitamin was masked for taste and flavor and was indistinguishable in consistency, appearance and taste from the control syrup containing the multivitamin only. The micronutrient supplements were prepared by Acme Laboratories, Dhaka Bangladesh. The experimental group received the zinc syrup containing the multivitamin (the vitamins were given at twice the recommended dietary allowance) in 2 divided doses daily for 2 weeks starting from the day of admission. The comparison group received the same multivitamin syrup alone. All the subjects received pivmecillinum in a dose of 60 mg/kg/day in 4 divided doses for 5 days. In both groups of patients, diarrhea subsided within 3-5 days. During hospitalization all the study children received a standard hospital diet of 100-125 kcal and 3-5 g protein per kg body weight daily in mixed food. When discharged at day-7, their mothers were given the bottles of syrup and were instructed to feed the child with the supplement daily at home for rest 7 days. On the 14th day, a health assistant visited the household, measured the amount of syrup taken and also enquired the mothers about any problems encountered during feeding of syrups. Children were followed up fortnightly for up to 6 months after the onset of diarrhoea to assess morbidity and growth. The following was investigated during the study period -Clinical evaluation: duration of illness, presence of blood in stool, tenesmus, and weight changes.Assessment of growth and growth velocity: Measurements included weight, height, triceps skinfold thickness (TSF) using standard technique (WHO)28. These were done before supplementation and at discharge. After supplementation, children were measured every two weeks at home. Weights were obtained to the nearest 10 g using an electronic digital scale (Secca model 770, Sweden) standarised with 5 and 10 kg standard weights in everyday morning and evening. Recubent length was measured in children less than two years of age using a slide board infantometer (Harpenden, St. Albans, England). In older children, standing height was determined with a Stadiometer . Mean of two consecutive height measurements to the nearest 0.5 cm was recorded as the observe value. Measurements were compared to Median NCHS Standard. Health workers were extensively trained in anthropometric measurements, until minimum intra-individual and inter individual variation was attainted. Statistical Analysis:The data were checked daily at recording by the investigators, cleaned and then entered in microcomputer using SPSS/PC+ (Windows 10.0). Data analysis was performed using SPSS/PC+ (Windows 10.0) and EPI Info (Nutrition)version 3.2.2. The consistency check was done using logical programs. Student and paired t-tests were used when data were normally distributed and non- parametric Mann-Whitney U tests were used when the distribution were skewed. Time sequence of proportions of recovery was compared between two groups using Kaplan Meier survival analysis. Proportions were compared using chi-squared test. Repeated measure analyses of variance were also undertaken to evaluate the changes in weight gain and length gain over the follow-up periods. Statistical significance was accepted at 5 percent level.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 12-59 months
2. Moderate malnutrition (61-75% Weight / Age - NCHS Median)
3. Duration of diarrhoea of 5 days
4. Culture confirmed shigella spp in stool on enrolment

Exclusion Criteria:

1. Measles infection in the past six months
2. Presence of obvious systemic illnesses
3. Severe malnutrition
4. Residence in a location requiring a journey of>2 hour from the Dhaka Hospital of the ICDDR,B
5. Refusal to give consent

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56
Dates: Start 1999-01; Study Completion 2002-04

PRIMARY OUTCOMES:
Age
Sex
Weight
Body Mass index
Duration of diarrhoea before admission
Stool volume
Dehydration status

SECONDARY OUTCOMES:
In blood: total and differential WBC counts,C-reactive protein, albumin, serum electrolytes and creatinine concentration
Quantitation of luminal neutriphils
Immune response
Duration of recovery
Presence of blood and mucous in stool
Weight gain
Length gain
Episodes of illness during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Swapan Kumar Roy, MBBS, M.Sc, Ph. D, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh

REFERENCES:
- [Derived] Roy SK, Raqib R, Khatun W, Azim T, Chowdhury R, Fuchs GJ, Sack DA. Zinc supplementation in the management of shigellosis in malnourished children in Bangladesh. Eur J Clin Nutr. 2008 Jul;62(7):849-55. doi: 10.1038/sj.ejcn.1602795. Epub 2007 Jun 6. PMID 17554249